CLINICAL TRIAL: NCT00601484
Title: A PHASE 2, 16 WEEK, MULTICENTER, RANDOMIZED, DOUBLE BLIND PLACEBO CONTROLLED, PARALLEL GROUP PROOF OF CONCEPT STUDY EVALUATING THE EFFICACY AND SAFETY OF PF-04383119 FOR THE TREATMENT OF PAIN ASSOCIATED WITH INTERSTITIAL CYSTITIS
Brief Title: An Effectiveness and Safety Study of PF-04383119 for the Treatment of Pain in Interstitial Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091010; IC POC (Other: Alias Study Number)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Cystitis, Interstitial
Keywords: Painful Bladder Syndrome; monoclonal antibody
MeSH Terms: conditions — Cystitis, Interstitial | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: PF-04383119
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04383119 — PF-04383119 200 mcg/kg IV, single dose
  Arms: 1
Drug: Placebo — placebo IV, single dose
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether PF-04383119 is effective in the treatment of pain associated with interstitial cystitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults at least 18 years of age;
* Moderate to severe interstitial cystitis, with a mean pain intensity score above a pre-defined level.

Exclusion Criteria:

* Less than 6 months since onset of interstitial cystitis symptoms;
* History of recurrent urinary tract infections, or genitourinary cancer;
* History of hepatitis B, C or human immunodeficiency virus (HIV);
* Use of certain drugs given into the bladder up to 1 month prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-03-17 (Actual); Primary Completion 2009-04-15 (Actual); Study Completion 2009-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (34):
  - Pivotal Research Center, Peoria, Arizona
  - Urology Associates of Central California, Fresno, California
  - Citrus Valley Medical Research Inc., Glendora, California
  - SD Uro-Research, San Diego, California
  - Boulder Medical Center, Boulder, Colorado
  - Hartford Hospital, Urogynecology Division, Hartford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Connecticut Clinical Research Center, Urology Specialists PC, Middlebury, Connecticut
  - Waterbury Neurology, Middlebury, Connecticut
  - Connecticut Urological Research at Grove Hill, New Britain, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Timothy M. Barczak, MD, LLC, New London, Connecticut
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Metropolitan Urology, Jeffersonville, Indiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - Michigan Institute of Urology, Utica, Michigan
  - Barnes Jewish West County Hospital, St Louis, Missouri
  - Washington University, Division of Urologic Surgery, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Quality Clinical Research Inc, Omaha, Nebraska
  - The Arthur Smith Institute for Urology, New Hyde Park, New York
  - University of Rochester Medical Center, Rochester, New York
  - Alliance Urology Specialists, PA, Greensboro, North Carolina
  - Tri-State Urologic Services PSC, Inc. dba The Urology Group, Cincinnati, Ohio
  - Parkhurst Research Organization, LLC, Bethany, Oklahoma
  - Triangle Urological Associates, Pittsburgh, Pennsylvania
  - Matrix Research, LLC (Administrative Only), Greer, South Carolina
  - The Urology Group, Greer, South Carolina
  - Mobley Research Center, Houston, Texas
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington
  - Northside Internal Medicine, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091010&StudyName=An%20Effectiveness%20and%20Safety%20Study%20of%20PF-04383119%20for%20the%20Treatment%20of%20Pain%20in%20Interstitial%20Cystitis

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanezumab: A single dose of tanezumab (RN624 or PF-04383119) 200 microgram per kilogram (mcg/kg) of body weight intravenous infusion over 10 minutes on Day 1. Participants were followed up to Week 16.
- Placebo: A single dose of placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over 10 minutes on Day 1. Participants were followed up to Week 16.
Period: Overall Study
Arm/Group | Tanezumab | Placebo
Started | 34 | 31
Treated | 34 | 30
Completed | 29 | 23
Not Completed | 5 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 4 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Randomized, but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab | Placebo | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (13.9) | 46.4 (16.6) | 44.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Pain Score at Week 6
Description: Participants assessed their average interstitial cystitis pain intensity during the last 24 hours on an 11-point numeric rating scale (NRS) ranging from 0 (no interstitial cystitis pain) to 10 (worst possible interstitial cystitis pain); where higher scores indicated higher pain. The average daily pain score was calculated as the mean of the scores over the last 7 days prior to each assessment time point. Here, 'Number analyzed' = participants with available data for each specified category.
Time Frame: Baseline, Week 6
Population: Restricted Full Analysis Set(rFAS): All randomized participants who received at least 1 dose of treatment, completed at least 5 diary days during 7 days prior to randomization, had at least 1 diary day post-randomization, and who provided baseline and post-randomization primary efficacy data for 4 or more days within the predefined diary windows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale
  Baseline | 6.4 (1.39) | 5.9 (1.15)
  Change at Week 6: number analyzed (Participants) | 28 | 23
  Change at Week 6 | -2.3 (1.88) | -1.1 (1.49)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Analysis was based on analysis of covariance (ANCOVA) model with terms for treatment, age, gender, body mass index (BMI), baseline severity of pain and concomitant medications (amitriptyline, pentosan polysulfate sodium, hydroxyzine) use; Test type: Superiority or Other; Least squares (LS) mean difference = -1.36, 90% CI 2-sided [-2.203 to -0.510], Standard Error of Mean 0.503

2. Secondary Outcome: Change From Baseline in Average Daily Pain Score at Week 2, 4, 10 and 16
Description: Participants assessed their average interstitial cystitis pain intensity during the last 24 hours on an 11-point NRS ranging from 0 (no interstitial cystitis pain) to 10 (worst possible interstitial cystitis pain); where higher scores indicated higher pain. The average daily pain score was calculated as the mean of the scores over the last 7 days prior to each assessment time point.
Time Frame: Baseline, Week 2, 4, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale
  Change at Week 2: number analyzed (Participants) | 30 | 28
  Change at Week 2 | -1.5 (1.64) | -0.9 (1.15)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -2.1 (2.04) | -1.0 (1.44)
  Change at Week 10: number analyzed (Participants) | 28 | 23
  Change at Week 10 | -2.2 (1.93) | -1.4 (1.87)
  Change at Week 16: number analyzed (Participants) | 27 | 22
  Change at Week 16 | -1.9 (1.92) | -1.7 (1.77)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 2: Analysis was based on ANCOVA model with terms for treatment, age, gender, BMI, baseline severity of pain and concomitant medications (amitriptyline, pentosan polysulfate sodium, hydroxyzine) use; Test type: Superiority or Other; LS mean difference = -0.68, 90% CI 2-sided [-1.363 to 0.011], Standard Error of Mean 0.410
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 4: Analysis was based on ANCOVA model with terms for treatment, age, gender, BMI, baseline severity of pain and concomitant medications (amitriptyline, pentosan polysulfate sodium, hydroxyzine) use; Test type: Superiority or Other; LS mean difference = -1.13, 90% CI 2-sided [-1.969 to -0.297], Standard Error of Mean 0.498
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 10: Analysis was based on ANCOVA model with terms for treatment, age, gender, BMI, baseline severity of pain and concomitant medications (amitriptyline, pentosan polysulfate sodium, hydroxyzine) use; Test type: Superiority or Other; LS mean difference = -0.85, 90% CI 2-sided [-1.790 to 0.090], Standard Error of Mean 0.559
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 16: Analysis was based on ANCOVA model with terms for treatment, age, gender, BMI, baseline severity of pain and concomitant medications (amitriptyline, pentosan polysulfate sodium, hydroxyzine) use; Test type: Superiority or Other; LS mean difference = -0.45, 90% CI 2-sided [-1.356 to 0.457], Standard Error of Mean 0.538

3. Secondary Outcome: Percent Change From Baseline in Average Daily Pain Score at Week 2, 4, 6, 10 and 16
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percent change
  Change at Week 2: number analyzed (Participants) | 30 | 28
  Change at Week 2 | -23.2 (26.41) | -15.9 (19.64)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -33.3 (34.52) | -17.1 (24.73)
  Change at Week 6: number analyzed (Participants) | 28 | 23
  Change at Week 6 | -36.3 (29.10) | -18.3 (26.88)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -35.0 (32.47) | -23.5 (30.66)
  Change at Week 16: number analyzed (Participants) | 27 | 22
  Change at Week 16 | -29.5 (32.45) | -28.6 (30.16)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -8.68, 90% CI 2-sided [-19.954 to 2.601], Standard Error of Mean 6.727
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -17.74, 90% CI 2-sided [-31.948 to -3.523], Standard Error of Mean 8.470
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 6: Analysis was based on ANCOVA model with terms for treatment, age, gender, BMI, baseline severity of pain and concomitant medications (amitriptyline, pentosan polysulfate sodium, hydroxyzine) use; Test type: Superiority or Other; LS mean difference = -20.66, 90% CI 2-sided [-34.347 to -6.971], Standard Error of Mean 8.138
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -13.58, 90% CI 2-sided [-29.612 to 2.452], Standard Error of Mean 9.532
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -7.75, 90% CI 2-sided [-22.580 to 7.080], Standard Error of Mean 8.807

4. Secondary Outcome: Change From Baseline in O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) Score at Week 2, 4, 6, 10 and 16
Description: The ICSI contained 4 questions that measured symptom severity including urinary urgency, urinary frequency, nocturia and pain/burning/discomfort/pressure in the bladder. Each question in the ICSI was rated on a 0 (no symptoms) to 5 (severe symptoms) scale, with higher scores indicating greater symptom severity. The sum of the individual question ratings was the total score for the ICSI. Total score ranged from 0 (no symptoms) to 20 (severe symptoms), with higher score indicating greater symptom severity.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale
  Baseline | 13.8 (2.75) | 13.2 (3.08)
  Change at Week 2 | -2.8 (2.98) | -2.1 (2.52)
  Change at Week 4: number analyzed (Participants) | 31 | 21
  Change at Week 4 | -3.2 (3.28) | -1.9 (2.77)
  Change at Week 6: number analyzed (Participants) | 26 | 18
  Change at Week 6 | -2.9 (3.75) | -1.2 (3.30)
  Change at Week 10: number analyzed (Participants) | 26 | 21
  Change at Week 10 | -2.0 (2.71) | -2.1 (3.45)
  Change at Week 16: number analyzed (Participants) | 19 | 13
  Change at Week 16 | -3.0 (3.22) | -2.2 (2.76)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.56, 90% CI 2-sided [-1.768 to 0.650], Standard Error of Mean 0.721
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -1.21, 90% CI 2-sided [-2.723 to 0.297], Standard Error of Mean 0.898
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -1.47, 90% CI 2-sided [-3.682 to 0.752], Standard Error of Mean 1.311
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 0.54, 90% CI 2-sided [-1.110 to 2.198], Standard Error of Mean 0.980
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -0.99, 90% CI 2-sided [-2.904 to 0.922], Standard Error of Mean 1.114

5. Secondary Outcome: Percent Change From Baseline in O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) Score at Week 2, 4, 6, 10 and 16
Description: as for outcome 4
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: RFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percent change
  Change at Week 2 | -21.0 (21.07) | -16.3 (21.15)
  Change at Week 4: number analyzed (Participants) | 31 | 21
  Change at Week 4 | -23.2 (24.62) | -14.5 (23.46)
  Change at Week 6: number analyzed (Participants) | 26 | 18
  Change at Week 6 | -20.5 (28.12) | -9.3 (27.01)
  Change at Week 10: number analyzed (Participants) | 26 | 21
  Change at Week 10 | -14.1 (18.01) | -15.8 (28.79)
  Change at Week 16: number analyzed (Participants) | 19 | 13
  Change at Week 16 | -21.0 (22.00) | -15.5 (19.34)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -4.41, 90% CI 2-sided [-13.650 to 4.826], Standard Error of Mean 5.510
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -8.65, 90% CI 2-sided [-20.493 to 3.192], Standard Error of Mean 7.041
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -9.72, 90% CI 2-sided [-26.775 to 7.343], Standard Error of Mean 10.089
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 3.76, 90% CI 2-sided [-8.950 to 16.465], Standard Error of Mean 7.532
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -8.72, 90% CI 2-sided [-22.299 to 4.851], Standard Error of Mean 7.906

6. Secondary Outcome: Change From Baseline in Number of Micturitions Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: The micturition frequency per 24 hours was calculated from the sum of voluntary voids divided by the number of diary days over which they were collected.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
micturitions per 24 hours
  Baseline | 14.2 (3.81) | 13.0 (4.54)
  Change at Week 2 | -1.1 (1.84) | -1.0 (2.54)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -0.8 (2.23) | -0.5 (2.85)
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -0.3 (3.78) | -0.6 (3.08)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -0.7 (3.99) | -0.8 (3.05)
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -0.5 (2.42) | -0.9 (3.18)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = 0.24, 90% CI 2-sided [-0.776 to 1.265], Standard Error of Mean 0.609
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS Mean difference = -0.09, 90% CI 2-sided [-1.220 to 1.044], Standard Error of Mean 0.674
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = 0.57, 90% CI 2-sided [-1.124 to 2.269], Standard Error of Mean 1.009
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 0.27, 90% CI 2-sided [-1.441 to 1.988], Standard Error of Mean 1.019
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = 0.99, 90% CI 2-sided [-0.307 to 2.283], Standard Error of Mean 0.769

7. Secondary Outcome: Percent Change From Baseline in Number of Micturitions Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: as for outcome 6
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Median (Full Range); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percent change
  Change at Week 2 | -9.8 [-28.0 to 20.7] | -7.4 [-45.0 to 39.6]
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -8.5 [-31.3 to 34.2] | -0.1 [-40.6 to 56.4]
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -8.9 [-33.6 to 101.8] | -8.9 [-39.9 to 86.7]
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -14.9 [-35.5 to 80.9] | -9.5 [-35.9 to 69.8]
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -5.0 [-37.9 to 45.9] | -10.2 [-34.8 to 57.9]
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 2: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7]) as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -1.68, 90% CI 2-sided [-9.05 to 5.76]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 4: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7]) as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -2.78, 90% CI 2-sided [-12.65 to 4.24]
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 6: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7]) as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = 0.04, 90% CI 2-sided [-8.96 to 7.90]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 10: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7]) as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -1.38, 90% CI 2-sided [-11.57 to 8.28]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 16: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7]) as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = 3.97, 90% CI 2-sided [-6.82 to 13.02]

8. Secondary Outcome: Change From Baseline in Number of Nocturnal Micturitions Per Night at Week 2, 4, 6, 10 and 16
Description: The nocturnal frequency per night was calculated as the sum of voluntary voids that occurred during a night's sleep, divided by the number of nights over which this was collected.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: micturitions per night
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 26
micturitions per night
  Baseline | 7.1 (5.37) | 5.8 (5.52)
  Change at Week 2: number analyzed (Participants) | 27 | 25
  Change at Week 2 | -1.5 (4.22) | -0.6 (3.48)
  Change at Week 4: number analyzed (Participants) | 29 | 23
  Change at Week 4 | -1.6 (4.72) | -1.5 (4.99)
  Change at Week 6: number analyzed (Participants) | 27 | 21
  Change at Week 6 | -1.3 (3.36) | -2.1 (4.78)
  Change at Week 10: number analyzed (Participants) | 26 | 20
  Change at Week 10 | -1.6 (4.45) | -1.5 (4.95)
  Change at Week 16: number analyzed (Participants) | 26 | 21
  Change at Week 16 | 0.1 (4.31) | -1.6 (5.82)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.72, 90% CI 2-sided [-2.414 to 0.983], Standard Error of Mean 1.010
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = 0.42, 90% CI 2-sided [-1.548 to 2.384], Standard Error of Mean 1.169
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = 1.31, 90% CI 2-sided [-0.075 to 2.693], Standard Error of Mean 0.821
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.33, 90% CI 2-sided [-2.178 to 1.512], Standard Error of Mean 1.093
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS Mean difference = 2.07, 90% CI 2-sided [0.038 to 4.112], Standard Error of Mean 1.208

9. Secondary Outcome: Percent Change From Baseline in Number of Nocturnal Micturitions Per Night at Week 2, 4, 6, 10 and 16
Description: The nocturnal frequency per night was calculated as the sum of voluntary voids that occurred during a night's sleep, divided by the number of nights over which this was collected. Percent change from baseline was calculated for participants who reported greater than 0 episodes at baseline.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: as for outcome 8
Measure: Median (Full Range); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 29 | 24
percent change
  Change at Week 2: number analyzed (Participants) | 27 | 24
  Change at Week 2 | -8.8 [-100.0 to 114.3] | -14.6 [-58.8 to 850.0]
  Change at Week 4: number analyzed (Participants) | 29 | 22
  Change at Week 4 | -12.5 [-100.0 to 160.0] | -41.4 [-100.0 to 400.0]
  Change at Week 6: number analyzed (Participants) | 27 | 20
  Change at Week 6 | -17.7 [-95.0 to 166.7] | -29.2 [-88.0 to 271.4]
  Change at Week 10: number analyzed (Participants) | 26 | 19
  Change at Week 10 | -23.7 [-100.0 to 183.3] | -25.0 [-92.0 to 214.3]
  Change at Week 16: number analyzed (Participants) | 26 | 20
  Change at Week 16 | 0.0 [-82.4 to 333.3] | -40.0 [-100.0 to 228.6]
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Hodges-Lehman median difference = -6.41, 90% CI 2-sided [-33.33 to 18.68]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hodges-Lehman median difference = 15.83, 90% CI 2-sided [-14.12 to 41.18]
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; Hodges-Lehman median difference = 19.17, 90% CI 2-sided [0.00 to 38.10]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; Hodges-Lehman median difference = -0.71, 90% CI 2-sided [-30.95 to 32.73]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; Hodges-Lehman median difference = 34.89, 90% CI 2-sided [-4.57 to 70.00]

10. Secondary Outcome: Change From Baseline in Number of Incontinence Episodes Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: The incontinence episode frequency per 24 hours was calculated as the sum of any incontinence episodes occurring during the diary period when this was measured, divided by the number of days over which they were recorded.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
episodes per 24 hours
  Baseline | 0.7 (1.21) | 1.0 (1.98)
  Change at Week 2 | -1.4 (3.05) | -2.0 (4.23)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -1.6 (3.09) | -2.1 (4.83)
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -1.5 (2.99) | -2.4 (4.95)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -1.7 (3.00) | -2.1 (4.62)
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -1.6 (3.28) | -2.4 (4.94)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = 0.04, 90% CI 2-sided [-0.529 to 0.610], Standard Error of Mean 0.340
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -0.52, 90% CI 2-sided [-1.077 to 0.043], Standard Error of Mean 0.334
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.22, 90% CI 2-sided [-0.835 to 0.396], Standard Error of Mean 0.366
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.22, 90% CI 2-sided [-0.718 to 0.273], Standard Error of Mean 0.294
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -0.30, 90% CI 2-sided [-1.044 to 0.445], Standard Error of Mean 0.442

11. Secondary Outcome: Percent Change From Baseline in Number of Incontinence Episodes Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: The incontinence episode frequency per 24 hours was calculated as the sum of any incontinence episodes occurring during the diary period when this was measured, divided by the number of days over which they were recorded. Percent change from baseline was calculated for participants who reported greater than 0 episodes at baseline.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'overall number of participants analyzed' = participants evaluable and had data available for this outcome measure and 'Number analyzed' = participants with available data for each specified category.
Measure: Median (Full Range); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 14 | 9
percent change
  Change at Week 2 | -97.3 [-100.0 to -24.5] | -87.6 [-100.0 to -17.4]
  Change at Week 4: number analyzed (Participants) | 14 | 8
  Change at Week 4 | -82.5 [-100.0 to -31.5] | -68.6 [-100.0 to 57.2]
  Change at Week 6: number analyzed (Participants) | 13 | 8
  Change at Week 6 | -100.0 [-100.0 to -32.2] | -70.3 [-100.0 to 14.2]
  Change at Week 10: number analyzed (Participants) | 14 | 7
  Change at Week 10 | -96.6 [-100.0 to -48.7] | -74.3 [-100.0 to 5.0]
  Change at Week 16: number analyzed (Participants) | 14 | 7
  Change at Week 16 | -93.5 [-100.0 to -30.3] | -81.7 [-100.0 to -9.5]
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Hodges-Lehman median difference = -1.24, 90% CI 2-sided [-27.56 to 5.37]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hodges-Lehman median difference = -22.43, 90% CI 2-sided [-56.39 to 0.00]
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; Hodges-Lehman median difference = -16.00, 90% CI 2-sided [-40.44 to 0.00]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; Hodges-Lehman median difference = -14.18, 90% CI 2-sided [-50.71 to 0.00]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; Hodges-Lehman median difference = -8.61, 90% CI 2-sided [-36.87 to 4.64]

12. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition at Week 2, 4, 6, 10 and 16
Description: Mean voided volume per micturition was calculated as the total urine volume voided (resulting from a toilet [voluntary] void) during the diary period when this was measured, divided by the number of toilet voids over which this occurred.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: milliliter (mL)/micturition
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
milliliter (mL)/micturition
  Baseline | 149.9 (64.65) | 172.2 (67.85)
  Change at Week 2 | 5.4 (43.18) | 1.4 (41.87)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | 2.0 (36.56) | 2.6 (49.90)
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -4.0 (45.30) | -0.4 (46.31)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -7.4 (43.26) | -8.4 (43.07)
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -1.4 (50.61) | -5.6 (41.48)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = 5.10, 90% CI 2-sided [-15.852 to 26.044], Standard Error of Mean 12.495
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = 4.27, 90% CI 2-sided [-17.216 to 25.764], Standard Error of Mean 12.802
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -2.81, 90% CI 2-sided [-25.917 to 20.307], Standard Error of Mean 13.741
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.73, 90% CI 2-sided [-21.626 to 20.162], Standard Error of Mean 12.416
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = 10.51, 90% CI 2-sided [-13.858 to 34.868], Standard Error of Mean 14.469

13. Secondary Outcome: Percent Change From Baseline in Mean Voided Volume Per Micturition at Week 2, 4, 6, 10 and 16
Description: as for outcome 12
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percent change
  Change at Week 2 | 3.8 (24.55) | -0.1 (22.07)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | 0.3 (21.29) | -0.8 (28.54)
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -2.8 (21.58) | -2.3 (29.04)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -2.7 (26.92) | -8.8 (23.97)
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -1.5 (29.52) | -5.3 (23.03)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = 3.63, 90% CI 2-sided [-8.049 to 15.316], Standard Error of Mean 6.968
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = 3.19, 90% CI 2-sided [-9.153 to 15.533], Standard Error of Mean 7.353
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.94, 90% CI 2-sided [-13.806 to 11.932], Standard Error of Mean 7.651
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 6.79, 90% CI 2-sided [-5.901 to 19.486], Standard Error of Mean 7.543
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = 4.77, 90% CI 2-sided [-9.221 to 18.765], Standard Error of Mean 8.310

14. Secondary Outcome: Change From Baseline in Mean Interstitial Cystitis Pain Severity Per Urinary Event at Week 2, 4, 6, 10 and 16
Description: Mean interstitial cystitis pain severity per urinary event (toilet void, accidental urine loss, urgency episode) was calculated as the mean of all pain severities recorded during the diary period when these events were measured. For each urinary event (toilet void, accidental urine loss, urgency episode), participants marked their associated level of pain intensity (or pressure, aching, burning, discomfort) using an 11-point NRS ranging from 0 denoting none (no pain), and 10 denoting worst (pain as bad as you can imagine), where higher scores indicated higher pain. Total mean interstitial cystitis pain severity per urinary event score ranged from 0 (no pain) to 10 worst (pain as bad as you can imagine), where higher scores indicated more pain.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale
  Baseline | 5.4 (1.78) | 4.7 (1.18)
  Change at Week 2 | -1.4 (1.69) | -0.5 (1.13)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -1.7 (1.96) | -0.4 (1.30)
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -1.7 (2.07) | -0.2 (1.42)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -1.6 (2.17) | -0.4 (1.58)
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -1.3 (2.09) | -0.5 (1.60)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.86, 90% CI 2-sided [-1.546 to -0.182], Standard Error of Mean 0.407
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -1.38, 90% CI 2-sided [-2.196 to -0.570], Standard Error of Mean 0.484
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -1.30, 90% CI 2-sided [-2.204 to -0.388], Standard Error of Mean 0.540
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -1.10, 90% CI 2-sided [-2.032 to -0.172], Standard Error of Mean 0.553
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -1.02, 90% CI 2-sided [-1.878 to -0.152], Standard Error of Mean 0.512

15. Secondary Outcome: Percent Change From Baseline in Mean Interstitial Cystitis Pain Severity Per Urinary Event at Week 2, 4, 6, 10 and 16
Description: as for outcome 14
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here 'number analyzed' signifies those participants who were evaluable for each specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percent change
  Change at Week 2 | -26.2 (31.24) | -13.1 (26.06)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -32.5 (37.82) | -8.2 (29.58)
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -29.9 (37.29) | -5.2 (37.85)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -25.9 (44.02) | -7.0 (37.00)
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -23.0 (41.99) | -10.7 (38.13)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -16.24, 90% CI 2-sided [-29.757 to -2.718], Standard Error of Mean 8.064
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -27.96, 90% CI 2-sided [-44.846 to -11.075], Standard Error of Mean 10.059
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -25.72, 90% CI 2-sided [-45.079 to -6.369], Standard Error of Mean 11.508
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -19.56, 90% CI 2-sided [-40.017 to 0.902], Standard Error of Mean 12.157
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -21.90, 90% CI 2-sided [-40.633 to -3.171], Standard Error of Mean 11.124

16. Secondary Outcome: Change From Baseline in Urinary Urgency Episodes Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: The urinary urgency episode per 24 hours was calculated as the sum of any urgency episodes occurring during the diary period when this was measured, divided by the number of days over which they were recorded.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
episodes per 24 hours
  Baseline | 8.5 (4.88) | 8.7 (6.75)
  Change at Week 2 | -1.7 (3.49) | -0.4 (2.97)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -1.8 (2.95) | 0.1 (3.39)
  Change at Week 6: number analyzed (Participants) | 29 | 23
  Change at Week 6 | -1.9 (4.74) | -0.1 (3.88)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -1.4 (5.91) | -0.9 (4.31)
  Change at Week 16: number analyzed (Participants) | 28 | 22
  Change at Week 16 | -2.1 (4.84) | -0.7 (4.12)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -1.50, 90% CI 2-sided [-2.942 to -0.057], Standard Error of Mean 0.860
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -2.08, 90% CI 2-sided [-3.458 to -0.705], Standard Error of Mean 0.820
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -2.13, 90% CI 2-sided [-4.265 to -0.004], Standard Error of Mean 1.267
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -1.45, 90% CI 2-sided [-4.029 to 1.124], Standard Error of Mean 1.531
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -2.24, 90% CI 2-sided [-4.419 to -0.063], Standard Error of Mean 1.293

17. Secondary Outcome: Percent Change From Baseline in Urinary Urgency Episodes Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: The urinary urgency episode per 24 hours was calculated as the sum of any urgency episodes occurring during the diary period when this was measured, divided by the number of days over which they were recorded. Percent change from baseline was calculated for participants who reported greater than 0 episodes at baseline.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: as for outcome 8
Measure: Median (Full Range); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 27
percent change
  Change at Week 2 | -21.5 [-100.0 to 90.1] | -4.7 [-100.0 to 221.0]
  Change at Week 4: number analyzed (Participants) | 30 | 24
  Change at Week 4 | -22.9 [-100.0 to 49.4] | 0.8 [-100.0 to 248.7]
  Change at Week 6: number analyzed (Participants) | 28 | 22
  Change at Week 6 | -30.4 [-100.0 to 101.8] | -1.6 [-100.0 to 297.5]
  Change at Week 10: number analyzed (Participants) | 28 | 21
  Change at Week 10 | -19.5 [-100.0 to 196.3] | -4.8 [-100.0 to 242.3]
  Change at Week 16: number analyzed (Participants) | 27 | 22
  Change at Week 16 | -32.1 [-100.0 to 98.4] | -6.7 [-100.0 to 144.7]
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 2: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7] as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -7.93, 90% CI 2-sided [-27.32 to 11.32]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 4: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7] as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -17.90, 90% CI 2-sided [-42.04 to 4.37]
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Week 6: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7] as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -24.44, 90% CI 2-sided [-51.58 to 0.67]
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Week 10: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7] as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -7.50, 90% CI 2-sided [-41.71 to 17.33]
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; Week 16: Van elteren test was used to compare the percent change from baseline between tanezumab and placebo using baseline average daily pain score (moderate [4 to less than 7] or severe [greater than or equal to 7] as stratification variable; Test type: Superiority or Other; Hodges-Lehman median difference = -21.37, 90% CI 2-sided [-54.76 to 7.92]

18. Secondary Outcome: Change From Baseline in Average Sleep Disturbance Score Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: Average sleep disturbance score was calculated from the sleep disturbance experienced over the previous night. The average sleep disturbance score per night was determined from calculating the mean of all sleep disturbance scores in the 7 days prior to each assessment time point. Participants answered the following question: "Over the past 24 hours, how much did the symptoms that you associate with your interstitial cystitis disturb your sleep?" Participants responded on a 5-point scale ranging from 0 (not at all) to 4 (extremely); where higher scores indicated more sleep disturbance.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale
  Baseline | 2.3 (0.73) | 2.1 (0.78)
  Change at Week 2: number analyzed (Participants) | 30 | 28
  Change at Week 2 | -0.5 (0.64) | -0.3 (0.51)
  Change at Week 4: number analyzed (Participants) | 31 | 25
  Change at Week 4 | -0.7 (0.76) | -0.3 (0.75)
  Change at Week 6: number analyzed (Participants) | 28 | 23
  Change at Week 6 | -0.7 (0.73) | -0.4 (0.69)
  Change at Week 10: number analyzed (Participants) | 29 | 22
  Change at Week 10 | -0.7 (0.76) | -0.3 (0.86)
  Change at Week 16: number analyzed (Participants) | 27 | 22
  Change at Week 16 | -0.5 (0.68) | -0.5 (0.63)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.32, 90% CI 2-sided [-0.591 to -0.040], Standard Error of Mean 0.165
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -0.36, 90% CI 2-sided [-0.734 to 0.020], Standard Error of Mean 0.225
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.37, 90% CI 2-sided [-0.724 to -0.015], Standard Error of Mean 0.211
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.41, 90% CI 2-sided [-0.806 to -0.005], Standard Error of Mean 0.238
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -0.12, 90% CI 2-sided [-0.470 to 0.223], Standard Error of Mean 0.206

19. Secondary Outcome: Percent Change From Baseline in Average Sleep Disturbance Score Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: Average sleep disturbance score was calculated from the sleep disturbance experienced over the previous night. The average sleep disturbance score per night was determined from calculating the mean of all sleep disturbance scores in the 7 days prior to each assessment time point. Participants answered the following question: "Over the past 24 hours, how much did the symptoms that you associate with your interstitial cystitis disturb your sleep?" Participants responded on a 5-point scale ranging from 0 (not at all) to 4 (extremely); where higher scores indicated more sleep disturbance. Percent change from baseline was calculated for participants who reported greater than 0 score at baseline.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 27
percent change
  Change at Week 2: number analyzed (Participants) | 30 | 27
  Change at Week 2 | -23.7 (29.81) | -11.6 (28.42)
  Change at Week 4: number analyzed (Participants) | 31 | 24
  Change at Week 4 | -32.0 (38.58) | -15.5 (33.54)
  Change at Week 6: number analyzed (Participants) | 28 | 22
  Change at Week 6 | -33.8 (35.41) | -17.4 (29.31)
  Change at Week 10: number analyzed (Participants) | 29 | 21
  Change at Week 10 | -28.3 (35.62) | -11.2 (52.83)
  Change at Week 16: number analyzed (Participants) | 27 | 21
  Change at Week 16 | -26.7 (35.40) | -23.8 (30.31)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -15.34, 90% CI 2-sided [-29.468 to -1.209], Standard Error of Mean 8.425
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -16.97, 90% CI 2-sided [-35.608 to 1.665], Standard Error of Mean 11.102
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -18.04, 90% CI 2-sided [-35.476 to -0.613], Standard Error of Mean 10.358
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -19.48, 90% CI 2-sided [-42.418 to 3.460], Standard Error of Mean 13.631
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -9.16, 90% CI 2-sided [-26.174 to 7.849], Standard Error of Mean 10.097

20. Secondary Outcome: Change From Baseline in Average Pain Score Associated With Sexual Activity Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: The average pain score associated with sexual activity was determined from calculating the mean of sexual activity scores of 7 days prior to each assessment time point. Participants answered the following question: "Over the past 24 hours, how much pain did you experience during or after sexual activity?" Participants responded on a 5-point scale ranging from 0 (no pain) to 4 (extremely painful); where higher scores indicated higher pain.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale
  Baseline | 2.1 (1.03) | 1.4 (0.84)
  Change at Week 2: number analyzed (Participants) | 12 | 11
  Change at Week 2 | -0.7 (0.99) | -0.0 (0.51)
  Change at Week 4: number analyzed (Participants) | 12 | 9
  Change at Week 4 | -0.7 (0.98) | -0.4 (0.47)
  Change at Week 6: number analyzed (Participants) | 10 | 11
  Change at Week 6 | -0.7 (1.24) | -0.2 (0.50)
  Change at Week 10: number analyzed (Participants) | 12 | 7
  Change at Week 10 | -0.7 (1.40) | -0.6 (0.54)
  Change at Week 16: number analyzed (Participants) | 10 | 8
  Change at Week 16 | -0.9 (0.95) | -0.0 (0.88)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.68, 90% CI 2-sided [-1.394 to 0.030], Standard Error of Mean 0.404
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -0.34, 90% CI 2-sided [-1.149 to 0.468], Standard Error of Mean 0.454
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.64, 90% CI 2-sided [-1.443 to 0.156], Standard Error of Mean 0.449
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.06, 90% CI 2-sided [-1.046 to 0.931], Standard Error of Mean 0.546
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -0.64, 90% CI 2-sided [-1.876 to 0.592], Standard Error of Mean 0.673

21. Secondary Outcome: Percent Change From Baseline in Average Pain Score Associated With Sexual Activity Per 24 Hours at Week 2, 4, 6, 10 and 16
Description: The average pain score associated with sexual activity was determined from calculating the mean of sexual activity scores in the 7 days prior to each assessment time point. Participants answered the following question: "Over the past 24 hours, how much pain did you experience during or after sexual activity?" Participants responded on a 5-point scale ranging from 0 (no pain) to 4 (extremely painful); where higher scores indicated higher pain. Percent change from baseline was calculated for participants who reported greater than 0 score at baseline.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 11 | 9
percent change
  Change at Week 2 | -28.5 (36.20) | -8.0 (29.94)
  Change at Week 4: number analyzed (Participants) | 11 | 8
  Change at Week 4 | -35.4 (35.65) | -38.6 (43.33)
  Change at Week 6: number analyzed (Participants) | 8 | 9
  Change at Week 6 | -31.6 (54.20) | -9.3 (55.81)
  Change at Week 10: number analyzed (Participants) | 11 | 6
  Change at Week 10 | -19.4 (83.01) | -47.7 (33.81)
  Change at Week 16: number analyzed (Participants) | 9 | 5
  Change at Week 16 | -43.5 (38.21) | -19.4 (75.54)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -34.25, 90% CI 2-sided [-72.879 to 4.375], Standard Error of Mean 21.509
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -30.97, 90% CI 2-sided [-75.230 to 13.285], Standard Error of Mean 24.418
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -37.18, 90% CI 2-sided [-90.620 to 16.265], Standard Error of Mean 28.740
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 5.77, 90% CI 2-sided [-74.604 to 86.142], Standard Error of Mean 43.222
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -21.35, 90% CI 2-sided [-164.142 to 121.438], Standard Error of Mean 70.862

22. Secondary Outcome: Change From Baseline in Pelvic Pain and Urgency/Frequency (PUF) Total Score at Week 2, 4, 6, 10 and 16
Description: The pelvic pain and urgency/frequency (PUF) was a 12-item questionnaire used to measure the severity of symptoms and the degree to which participants were bothered. Symptom questions include 3, 4, or 5 ranked answers, with higher answers indicating more voids, or greater frequency of pain. The bother questions consisted of 4 ranked answers from 0-never to 3-always with higher answers indicating more bothering. Total score was calculated as the sum of symptom score and bother score and ranged from 0 (no symptoms/bother) to 35 (higher symptom severity/bother), where a higher score indicated greater symptom severity and higher bother from pelvic pain and frequency.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale
  Baseline | 22.8 (3.82) | 21.1 (3.91)
  Change at Week 2 | -4.0 (3.95) | -3.3 (4.59)
  Change at Week 4: number analyzed (Participants) | 31 | 21
  Change at Week 4 | -4.4 (5.43) | -3.0 (4.06)
  Change at Week 6: number analyzed (Participants) | 26 | 18
  Change at Week 6 | -5.0 (5.51) | -3.6 (4.49)
  Change at Week 10: number analyzed (Participants) | 26 | 21
  Change at Week 10 | -4.2 (4.87) | -3.5 (4.18)
  Change at Week 16: number analyzed (Participants) | 19 | 13
  Change at Week 16 | -4.3 (5.81) | -3.6 (2.96)

23. Secondary Outcome: Percent Change From Baseline in Pelvic Pain and Urgency/Frequency (PUF) Symptom Total Score at Week 2, 4, 6, 10 and 16
Description: The pelvic pain and urgency/frequency (PUF) was a 12-item questionnaire used to measure the severity of symptoms and the degree to which participants were bothered. Symptom questions include 3, 4, or 5 ranked answers, with higher answers indicating more voids, or greater frequency of pain. The bother questions each of 4 ranked answers from 0-never, to 3-always with higher answers indicating more bothering. Total score was calculated as the sum of symptom score and bother score and ranged from 0 (no symptoms/bother) to 35 (higher symptom severity/bother), where a higher score indicated greater symptom severity and higher bother from pelvic pain and frequency.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percent change
  Change at Week 2 | -17.0 (16.23) | -15.6 (21.67)
  Change at Week 4: number analyzed (Participants) | 31 | 21
  Change at Week 4 | -18.9 (24.33) | -14.9 (19.52)
  Change at Week 6: number analyzed (Participants) | 26 | 18
  Change at Week 6 | -21.4 (23.14) | -18.5 (22.38)
  Change at Week 10: number analyzed (Participants) | 26 | 21
  Change at Week 10 | -17.8 (20.49) | -17.3 (20.67)
  Change at Week 16: number analyzed (Participants) | 19 | 13
  Change at Week 16 | -17.9 (23.81) | -18.3 (14.98)

24. Secondary Outcome: Change From Baseline in O'Leary-Sant Interstitial Cystitis Problem Index (ICPI) Score at Week 2, 4, 6, 10 and 16
Description: The ICPI contained 4 questions that measured how problematic the symptoms (urinary urgency, urinary frequency, nocturnal and pain/burning/discomfort/pressure in the bladder) were for the participant. Each question in the ICPI was rated on a 0-4 scale, where 0= no problem and 4= big problem. The sum of the individual question ratings was the total score for the ICPI. Total score ranged from 0 (no problem) to 16 (big problem), with higher score indicating greater problematic symptom.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale
  Baseline | 12.3 (2.25) | 11.7 (2.52)
  Change at Week 2 | -3.1 (3.02) | -1.8 (2.54)
  Change at Week 4: number analyzed (Participants) | 31 | 21
  Change at Week 4 | -3.3 (3.71) | -2.1 (2.60)
  Change at Week 6: number analyzed (Participants) | 26 | 18
  Change at Week 6 | -3.2 (3.53) | -2.1 (2.80)
  Change at Week 10: number analyzed (Participants) | 26 | 21
  Change at Week 10 | -2.5 (2.23) | -2.5 (2.71)
  Change at Week 16: number analyzed (Participants) | 19 | 13
  Change at Week 16 | -2.8 (2.62) | -2.3 (3.25)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -1.24, 90% CI 2-sided [-2.562 to 0.081], Standard Error of Mean 0.788
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -1.12, 90% CI 2-sided [-2.782 to 0.535], Standard Error of Mean 0.986
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -1.11, 90% CI 2-sided [-3.036 to 0.819], Standard Error of Mean 1.140
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.16, 90% CI 2-sided [-1.534 to 1.221], Standard Error of Mean 0.816
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -0.54, 90% CI 2-sided [-2.398 to 1.320], Standard Error of Mean 1.083

25. Secondary Outcome: Percent Change From Baseline in O'Leary-Sant Interstitial Cystitis Problem Index (ICPI) Score Week 2, 4, 6, 10 and 16
Description: The ICPI contained 4 questions that measured how problematic the symptoms (urinary urgency, urinary frequency, nocturia and pain/burning/discomfort/pressure in the bladder) were for the participant. Each question in the ICPI was rated on a 0-4 scale, where 0= no problem and 4= big problem. The sum of the individual question ratings was the total score for the ICPI. Total score ranged from 0 (no problem) to 16 (big problem), with higher score indicating greater problematic symptom.
Time Frame: Baseline, Week 2, 4, 6, 10, 16
Population: rFAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percent change
  Change at Week 2 | -26.0 (26.02) | -14.6 (21.65)
  Change at Week 4: number analyzed (Participants) | 31 | 21
  Change at Week 4 | -27.2 (32.99) | -18.3 (22.88)
  Change at Week 6: number analyzed (Participants) | 26 | 18
  Change at Week 6 | -26.4 (30.04) | -18.6 (25.30)
  Change at Week 10: number analyzed (Participants) | 26 | 21
  Change at Week 10 | -21.2 (21.68) | -23.0 (25.21)
  Change at Week 16: number analyzed (Participants) | 19 | 13
  Change at Week 16 | -24.6 (25.00) | -18.3 (26.07)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean difference = -10.99, 90% CI 2-sided [-22.250 to 0.277], Standard Error of Mean 6.718
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -8.43, 90% CI 2-sided [-23.001 to 6.132], Standard Error of Mean 8.660
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; LS mean difference = -8.14, 90% CI 2-sided [-24.602 to 8.327], Standard Error of Mean 9.737
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -1.45, 90% CI 2-sided [-13.948 to 11.040], Standard Error of Mean 7.406
Statistical Analysis 5: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; LS mean difference = -7.83, 90% CI 2-sided [-23.884 to 8.234], Standard Error of Mean 9.352

26. Secondary Outcome: Number of Participants With Global Response Assessment (GRA) at Weeks 6, and 16
Description: Participants were asked the following question: "Compared to when you began this trial, how would you rate your interstitial cystitis symptoms now?" Participants responded on a 7-point symmetric scale where 1 = markedly worse, 2 = moderately worse, 3 = slightly worse, 4 = no change, 5 = slightly improved, 6 = moderately improved and 7 = markedly improved; where higher scores indicated improvement. Participants who responded as 6 (moderately improved) or 7 (markedly improved) were defined as treatment responders. Number of participants with response based on GRA scale for all scale categories were reported in this outcome measure.
Time Frame: Week 6, 16
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 17
Participants
  Week 6: Markedly worse | 0 | 1
  Week 6: Moderately worse | 1 | 0
  Week 6: Slightly worse | 2 | 3
  Week 6: No change | 5 | 6
  Week 6: Slightly improved | 7 | 5
  Week 6: Moderately improved | 5 | 1
  Week 6: Markedly improved | 5 | 1
  Week 16: Moderately worse: number analyzed (Participants) | 19 | 13
  Week 16: Moderately worse | 2 | 1
  Week 16: Slightly worse: number analyzed (Participants) | 19 | 13
  Week 16: Slightly worse | 1 | 0
  Week 16: No change: number analyzed (Participants) | 19 | 13
  Week 16: No change | 5 | 5
  Week 16: Slightly improved: number analyzed (Participants) | 19 | 13
  Week 16: Slightly improved | 2 | 5
  Week 16: Moderately improved: number analyzed (Participants) | 19 | 13
  Week 16: Moderately improved | 5 | 2
  Week 16: Markedly improved: number analyzed (Participants) | 19 | 13
  Week 16: Markedly improved | 4 | 0
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 6: Analysis was based on proportional odds analysis, to determine the odds ratio for the odds of responding (compared to not responding) on Tanezumab vs placebo; Test type: Superiority or Other; Odds Ratio (OR) = 5.064, 90% CI 2-sided [1.709 to 15.007]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 16: Analysis was based on proportional odds analysis, to determine the odds ratio for the odds of responding (compared to not responding) on Tanezumab vs placebo; Test type: Superiority or Other; Odds Ratio (OR) = 2.722, 90% CI 2-sided [0.756 to 9.795]

27. Secondary Outcome: Patient's Global Satisfaction Assessment
Description: Participant global satisfaction was assessed using Patient Reported Treatment Impact (PRTI) which is a self-administered questionnaire containing 4 items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participants were asked the following question: "Overall, how satisfied are you with the drug that you received since you entered this trial?" Participant's response was rated on a 5-point scale where 1=extremely dissatisfied (dissatisfy), 2=dissatisfied, 3=neither satisfied nor dissatisfied (satisfy/dissatisfy), 4=satisfied and 5=extremely satisfied; where higher scores indicated more satisfaction. Number of participants with each response was reported in this outcome measure.
Time Frame: Week 6, 16
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 16
Participants
  Week 6: Extremely satisfied | 5 | 0
  Week 6: Satisfied | 7 | 6
  Week 6:Neither satisfied nor dissatisfied | 7 | 4
  Week 6: Dissatisfied | 4 | 4
  Week 6: Extremely dissatisfied | 2 | 2
  Week 16: Extremely satisfied: number analyzed (Participants) | 19 | 13
  Week 16: Extremely satisfied | 4 | 1
  Week 16: Satisfied: number analyzed (Participants) | 19 | 13
  Week 16: Satisfied | 7 | 6
  Week16:Neither satisfied nor dissatisfied: number analyzed (Participants) | 19 | 13
  Week16:Neither satisfied nor dissatisfied | 5 | 2
  Week 16: Dissatisfied: number analyzed (Participants) | 19 | 13
  Week 16: Dissatisfied | 2 | 2
  Week 16: Extremely dissatisfied: number analyzed (Participants) | 19 | 13
  Week 16: Extremely dissatisfied | 1 | 2

28. Secondary Outcome: Patient's Global Preference Assessment at Weeks 6, and 16
Description: Participant global preference was assessed using PRTI which is self-administered questionnaire containing 4 items to assess participant satisfaction, previous treatment, preference and willingness to continue using study medication. Participant reported previous treatment under following categories: lifestyle interventions, physical therapies, toileting programs, drug given into bladder, drug taken by mouth, surgery and no treatment. Participants' preference was assessed using following categories: definitely prefer current drug, slightly prefer current drug, no preference, definitely prefer prior treatment and slightly prefer prior treatment. Number of participants under each of the categories was reported in this outcome measure. For previous treatment, a single participant may be represented in more than 1 category.
Time Frame: Week 6, 16
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 16
Participants
  Week 6: Lifestyle interventions | 10 | 5
  Week 6: Physical therapies | 6 | 1
  Week 6: Toileting programs | 1 | 0
  Week 6: Drug given into bladder | 8 | 4
  Week 6: Drug taken by mouth | 18 | 10
  Week 6: Surgery | 2 | 2
  Week 6: No Treatment | 6 | 2
  Week 6: Definitely prefer current drug | 9 | 2
  Week 6: Slightly prefer current drug | 4 | 4
  Week 6: No preference | 9 | 5
  Week 6: Definitely prefer prior treatment | 3 | 5
  Week 16: Lifestyle interventions: number analyzed (Participants) | 19 | 13
  Week 16: Lifestyle interventions | 10 | 5
  Week 16: Physical therapies: number analyzed (Participants) | 19 | 13
  Week 16: Physical therapies | 5 | 0
  Week 16: Toileting programs: number analyzed (Participants) | 19 | 13
  Week 16: Toileting programs | 2 | 0
  Week 16: Drug given into bladder: number analyzed (Participants) | 19 | 13
  Week 16: Drug given into bladder | 7 | 2
  Week 16: Drug taken by mouth: number analyzed (Participants) | 19 | 13
  Week 16: Drug taken by mouth | 15 | 10
  Week 16: Surgery: number analyzed (Participants) | 19 | 13
  Week 16: Surgery | 3 | 3
  Week 16: No Treatment: number analyzed (Participants) | 19 | 13
  Week 16: No Treatment | 2 | 1
  Week16: Definitely prefer current drug: number analyzed (Participants) | 19 | 13
  Week16: Definitely prefer current drug | 6 | 1
  Week 16: Slightly prefer current drug: number analyzed (Participants) | 19 | 13
  Week 16: Slightly prefer current drug | 5 | 4
  Week 16: No preference: number analyzed (Participants) | 19 | 13
  Week 16: No preference | 4 | 3
  Week 16: Slightly prefer prior treatment: number analyzed (Participants) | 19 | 13
  Week 16: Slightly prefer prior treatment | 1 | 0
  Week16: Definitely prefer prior treatment: number analyzed (Participants) | 19 | 13
  Week16: Definitely prefer prior treatment | 3 | 5

29. Secondary Outcome: Patient Willingness to Re-use Medicine Assessment
Description: Participant willingness to re-use study medication was assessed using PRTI which is a self-administered questionnaire containing 4 items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participants were asked the following question: "In the future, would you be willing to use the same drug that you have received since you entered this trial for your interstitial cystitis?" Participant willingness to re-use study medication was assessed using following categories: definitely want to re-use, might want to re-use, not sure, might not want to re-use, and definitely would not want to re-use.
Time Frame: Week 6, 16
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 16
Participants
  Week 6: Definitely want to re-use | 9 | 3
  Week 6: Might want to re-use | 5 | 5
  Week 6: Not sure | 9 | 3
  Week 6: Might not want to re-use | 0 | 1
  Week 6: Definitely not want to re-use | 2 | 4
  Week 16: Definitely want to re-use: number analyzed (Participants) | 19 | 13
  Week 16: Definitely want to re-use | 7 | 4
  Week 16: Might want to re-use: number analyzed (Participants) | 19 | 13
  Week 16: Might want to re-use | 5 | 3
  Week 16: Not sure: number analyzed (Participants) | 19 | 13
  Week 16: Not sure | 2 | 1
  Week 16: Might not want to re-use: number analyzed (Participants) | 19 | 13
  Week 16: Might not want to re-use | 3 | 2
  Week 16:Definitely not want re-use: number analyzed (Participants) | 19 | 13
  Week 16:Definitely not want re-use | 2 | 3

30. Secondary Outcome: Percentage of Participants Who Use Rescue Medication
Description: In case of inadequate pain relief or worsening symptoms of interstitial cystitis, any United States Food and Drug Administration (US FDA) approved commercial product of acetaminophen 500 milligram (mg) tablet/capsule could be taken as rescue medication.
Time Frame: Baseline up to Week 16
Population: rFAS population: all randomized participants who received at least 1 dose of treatment, completed at least 5 diary days during 7 days prior to randomization, had at least 1 diary day post-randomization, and who provided baseline and post-randomization primary efficacy data for 4 or more days within the predefined diary windows.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
percentage of participants | 48.4 | 46.4

31. Secondary Outcome: Ratio of Number of Days Rescue Medication Used
Description: In case of inadequate pain relief or worsening symptoms of interstitial cystitis, any US FDA approved commercial product of acetaminophen 500 mg tablet/capsule could be taken as rescue medication. Results were normalized by days rescue medication was used relative to the total number of days participant was in the study.
Time Frame: Baseline up to Week 16
Population: as for outcome 30
Measure: Median (Full Range); unit: ratio
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
ratio | 0.00 [0.0 to 0.6] | 0.00 [0.0 to 0.7]

32. Secondary Outcome: Average Number of Doses Per Day of Rescue Medication Used
Description: In case of inadequate pain relief or worsening symptoms of interstitial cystitis, any US FDA approved commercial product of acetaminophen 500 mg tablet/capsule could be taken as rescue medication. Results were normalized by doses of rescue medication used relative to the total number of days participant was in the study.
Time Frame: Baseline up to Week 16
Population: as for outcome 30
Measure: Median (Full Range); unit: doses per day
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
doses per day | 0.00 [0.0 to 1.7] | 0.00 [0.0 to 0.9]

33. Secondary Outcome: Amount of Rescue Medication Taken Per Day
Description: In case of inadequate pain relief or worsening symptoms of interstitial cystitis, any US FDA approved commercial product of acetaminophen 500 mg tablet/capsule could be taken as rescue medication. Results were normalized by amount of rescue medication (in mg) relative to the total number of days participant was in the study.
Time Frame: Baseline up to Week 16
Population: as for outcome 30
Measure: Median (Full Range); unit: mg per day
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
mg per day | 0.00 [0.0 to 1657.1] | 0.00 [0.0 to 724.0]

34. Secondary Outcome: Time to First Dose of Rescue Medication as a Proportion of Total Days in Study
Description: In case of inadequate pain relief or worsening symptoms of interstitial cystitis, any US FDA approved commercial product of acetaminophen 500 mg tablet/capsule could be taken as rescue medication. Time to first dose of rescue medication was defined as the time (in days) from the first dose of study drug to the time of first dose of rescue medication use. Results were normalized by days (time [in days] to first dose of rescue medication) relative to the total number of days participant was in the study and reported in terms of proportion of total days in study.
Time Frame: Baseline up to Week 16
Population: as for outcome 30
Measure: Median (Full Range); unit: proportion of days
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 31 | 28
proportion of days | 0.00 [0.0 to 0.9] | 0.00 [0.0 to 1.0]

35. Secondary Outcome: Plasma and Urine Total Nerve Growth Factor (NGF) Concentration
Description: Plasma Total NGF levels were assayed using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. Urine NGF was not analyzed because no reliable assay method was available for assessing urine NGF.
Time Frame: Day 1 (1 hour pre-dose), Week 2, 4, 6, 10, 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
  Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 25
picogram per milliliter (pg/mL)
  Day 1 (pre-dose) | 16.47 (7.38) | 16.70 (7.33)
  Week 2: number analyzed (Participants) | 29 | 22
  Week 2 | 1943.45 (579.77) | 17.13 (7.88)
  Week 4: number analyzed (Participants) | 29 | 21
  Week 4 | 2654.76 (913.40) | 17.34 (4.86)
  Week 6: number analyzed (Participants) | 25 | 23
  Week 6 | 2542.80 (926.78) | 16.49 (8.64)
  Week 10: number analyzed (Participants) | 23 | 22
  Week 10 | 2396.09 (861.74) | 13.63 (6.69)
  Week 16: number analyzed (Participants) | 27 | 22
  Week 16 | 2202.04 (1014.21) | 15.47 (7.89)

36. Secondary Outcome: Heparin-binding Epidermal Growth Factor-like Growth Factor (HB-EGF) Urine Concentration
Description: HB-EGF urine concentration (in picogram per milliliter [pg/mL]) at specified time points is reported here.
Time Frame: Day 1 (1 hour pre-dose), Week 2, 4, 6, 10, 16
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 32 | 26
pg/mL
  Day 1 (pre-dose): number analyzed (Participants) | 32 | 24
  Day 1 (pre-dose) | 108.70 (71.15) | 114.05 (81.68)
  Week 2: number analyzed (Participants) | 31 | 26
  Week 2 | 126.08 (48.30) | 109.48 (61.93)
  Week 4: number analyzed (Participants) | 32 | 22
  Week 4 | 123.59 (73.19) | 120.09 (62.51)
  Week 6: number analyzed (Participants) | 30 | 24
  Week 6 | 119.54 (80.83) | 114.84 (59.03)
  Week 10: number analyzed (Participants) | 28 | 21
  Week 10 | 100.94 (60.87) | 115.39 (65.66)
  Week 16: number analyzed (Participants) | 29 | 23
  Week 16 | 115.72 (55.14) | 128.60 (75.62)

37. Secondary Outcome: Anti-Proliferative Factor (APF) Urine Concentration
Description: APF activity was determined using 3 H-thymidine incorporation assay. The results were expressed as the percentage of inhibition of 3 H-thymidine incorporation in epithelial cells from urine specimens in the presence of anti proliferative factor.
Time Frame: Day 1 (1 hour pre-dose), Week 2, 4, 6, 10, 16
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 32 | 27
percentage of inhibition
  Day 1 (pre-dose): number analyzed (Participants) | 32 | 26
  Day 1 (pre-dose) | 141.40 (43.33) | 157.87 (76.65)
  Week 2: number analyzed (Participants) | 31 | 27
  Week 2 | 157.66 (70.74) | 156.96 (54.68)
  Week 4: number analyzed (Participants) | 32 | 22
  Week 4 | 146.25 (39.04) | 163.80 (72.75)
  Week 6: number analyzed (Participants) | 30 | 24
  Week 6 | 161.38 (54.52) | 149.07 (32.81)
  Week 10: number analyzed (Participants) | 28 | 21
  Week 10 | 144.58 (55.21) | 162.45 (62.07)
  Week 16: number analyzed (Participants) | 29 | 23
  Week 16 | 152.55 (56.72) | 163.02 (59.98)

38. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination
Description: Physical examination included the examination of general appearance, skin, neck, eyes, ears, nose, throat, cardiovascular assessment including rhythm, and presence of other cardiac abnormalities (for example gallops, murmurs, cardiomegaly), respiratory system, gastrointestinal system, genitourinary system, musculoskeletal system and any additional assessments necessary to establish baseline status. Clinically significant change in physical examination was based on investigator's discretion.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 34 | 30
Participants | 0 | 0

39. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included the assessment of the following: body temperature, blood pressure, heart rate and respiratory rate. Clinically significant change in vital signs was based on investigator's discretion.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 34 | 30
Participants | 0 | 0

40. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Body Weight
Description: Clinically significant change in body weight was based on investigator's discretion.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 34 | 30
Participants | 0 | 0

41. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Neurologic Examination
Description: Neurological examination included the assessment of cranial nerve function, coordination, reflexes, mental state, motor function, proprioception, gait and station, and sensory function (sharp sensation, warm/cold sensation, light touch, deep pressure, and vibration sensation). Clinically significant change in neurologic examination was based on investigator's discretion.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 3 | 2

42. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG)
Description: Clinically significant criteria for ECG abnormality: PR interval (maximum increase from Baseline of >=25% [only if Baseline value was greater than 200 millisecond] or otherwise 50%), QRS complex (maximum increase from Baseline of >=25% [only if Baseline value was greater than 200 millisecond] or otherwise 50%), QT interval, QT interval corrected using the Fridericia's formula (QTcF) (maximum increase from Baseline of >= 30 to <60; or >=60), QT interval corrected using the Bazett's formula (QTcB) (maximum increase from Baseline of >= 30 to <60; or >=60) and RR interval.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 34 | 29
Participants
  PR interval (maximum increase from Baseline of >=25 or 50%) | 0 | 0
  QRS complex (maximum increase from Baseline of >=25 or 50%) | 0 | 0
  QTcB (maximum increase from Baseline of >= 30 to <60) | 4 | 2
  QTcB (maximum increase from Baseline of >=60) | 0 | 0
  QTcF (maximum increase from Baseline of >= 30 to <60) | 0 | 0
  QTcF (maximum increase from Baseline of >=60) | 0 | 0

43. Secondary Outcome: Post-void Residual (PVR) Volume
Description: PVR volume is an objective assessment of the amount of urine (in milliliter) left in the bladder after normal urination and monitored whether the active treatment had an adverse effect on lower urinary tract voiding function. The PVR volume was assessed using trans-abdominal ultrasound (for example, bladder scanner) with the participant in a supine position immediately after voluntary urination.
Time Frame: Baseline, Week 2, 6, 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 34 | 30
milliliter
  Baseline | 28.8 (32.68) | 40.2 (48.25)
  Week 2: number analyzed (Participants) | 32 | 28
  Week 2 | 25.9 (34.24) | 33.5 (48.62)
  Week 6: number analyzed (Participants) | 29 | 23
  Week 6 | 34.4 (35.26) | 38.6 (61.56)
  Week 16: number analyzed (Participants) | 28 | 25
  Week 16 | 49.4 (56.82) | 21.8 (38.81)

44. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory abnormalities: Hematology parameters: red blood cell count: <0.8*lower limit of normal (LLN); reticulocytes count (absolute or percent): <0.5*LLN or greater than (>) 1.5*upper limit of normal (ULN); Platelets: <0.5*LLN or >1.75*ULN; white blood cell count: <0.6*LLN or >1.5*ULN; neutrophils (absolute or percent): <0.8*LLN or >1.2*ULN; basophils (absolute or percent): >1.2*ULN; lymphocytes (absolute or percent): <0.8*LLN or >1.2*ULN; monocytes (absolute or percent): >1.2*ULN. Serum Chemistry parameters: sodium: <0.95*LLN or >1.05*ULN, potassium, chloride, bicarbonate, calcium: <0.9*LLN or >1.1*ULN; magnesium: >1.1*ULN or <0.9*LLN; BUN (blood urea nitrogen): >1.3* ULN, creatinine: >1.3*ULN; aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase : >3.0*ULN ; total bilirubin: >1.5*ULN; albumin: <0.8*LLN or >1.2*ULN and glucose: <0.6*LLN or >1.5*ULN.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 23 | 18

45. Secondary Outcome: Number of Participants With Presence of Anti-Drug Antibody (ADA)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using a semi quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1, Week 4, 6, 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab
Number analyzed (Participants) | 32
Participants
  Day 1: number analyzed (Participants) | 31
  Day 1 | 0
  Week 4 | 0
  Week 6: number analyzed (Participants) | 30
  Week 6 | 0
  Week 16: number analyzed (Participants) | 28
  Week 16 | 0

46. Secondary Outcome: Plasma Concentration of Tanezumab
Time Frame: 0 hour (pre-dose), 1, 2 hours post-dose on Day 1; and at Week 2, 4, 6, 10, 16
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tanezumab
Number analyzed (Participants) | 32
nanogram per milliliter (ng/mL)
  Day 1 0 hour pre-dose | 82.25 (435.80)
  Day 1 1 hour post-dose | 6070.81 (2521.35)
  Day 1 2 hour post-dose: number analyzed (Participants) | 30
  Day 1 2 hour post-dose | 5520.63 (1558.81)
  Week 2: number analyzed (Participants) | 29
  Week 2 | 1885.34 (403.93)
  Week 4 | 1214.59 (410.16)
  Week 6: number analyzed (Participants) | 30
  Week 6 | 888.70 (311.17)
  Week 10: number analyzed (Participants) | 25
  Week 10 | 338.10 (144.84)
  Week 16: number analyzed (Participants) | 28
  Week 16 | 104.07 (99.37)

ADVERSE EVENTS:
Description: The same event may appear as both an Adverse Event and a Serious Adverse Event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Analysis performed on safety analysis set.
Arm/Group | Tanezumab | Placebo
Serious Adverse Events (participants affected / at risk) | 2/34 | 4/30
Other Adverse Events (participants affected / at risk) | 23/34 | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=34) | Placebo (N=30)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=34) | Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Altered visual depth perception (Eye disorders) | 1 | 0
Blepharospasm (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 0
Feeling hot (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 1
Irritability (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2
Herpes simplex (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Formication (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 5
Hyperaesthesia (Nervous system disorders) | 3 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 6 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1
Tongue paralysis (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Perineal cyst (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Endodontic procedure (Surgical and medical procedures) | 1 | 0
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.